CLINICAL TRIAL: NCT07135024
Title: Prospective Register Study to Assess Eligibility for and Efficacy of Surgical Treatment in Patients With nEuRovascular Conflict
Acronym: PETER registry
Status: Not yet recruiting | Type: Observational
Sponsor: Gerrit A Schubert (Other)
Collaborators: NeuroResearchOffice at Cantonal Hospital Aarau (Unknown)
Responsible Party: Sponsor-Investigator, Gerrit A Schubert, Head of Neurosurgery, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Other Study IDs: PETER registry
Record Dates: First submitted 2025-08-05; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Trigeminal Neuralgia; Tic Douloureux; Facial Pain; Glossopharyngeal Neuralgia; Hemifacial Spasm; Neurovascular Conflict
Keywords: Trigeminal Neuralgia; Registry; prospective study; eligibility determination; efficacy, treatment; Follow-Up Studies; indication; microvascular decompression; Jannetta; tic douloureux; hemifacial spasm; neurovascular conflict; glossopharyngeal neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia; Facial Pain; Glossopharyngeal Nerve Diseases; Hemifacial Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the registry is a multicenter, prospective long-term data collection of patients suspected neurovascular conflict and referred for possible microvascular decompression (Jannetta procedure). The registry relies exclusively on routinely collected clinical data, which are gathered in a standardized and privacy-compliant manner as part of everyday clinical practice. By systematically compiling this information across multiple centers, valuable insights into the effectiveness, potential side effects, and long-term outcomes of this surgical treatment can be gained. The registry will serve as a foundation for future scientific analyses and is intended to help answer relevant research questions regarding the treatment of trigeminal neuralgia based on solid evidence.

ELIGIBILITY:
Inclusion Criteria:

* suspected neurovascular conflict
* signed consent for further use of routine clinical data as accepted by local regulations

Exclusion Criteria:

* refusal of further use of routine clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohort will be selected from local Department of Neurosurgery of participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 5001 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief after surgical treatment | From enrolment to last follow-up 5 yrs after surgery
  Efficacy of microvascular decompression surgery, defined by the change in pain as assessed by the patient using the Visual Analog Scale (VAS) from 0 to 100 mm, with higher scores representing worse outcomes.
Face specific pain relief after surgical treatment | From enrolment to last follow-up 5 yrs after surgery
  Efficacy of microvascular decompression surgery, defined by the change in facial pain and pain interference as assessed by the patient using the Brief Pain Inventory-Facial (BPI-Facial), with numerical scores ranging from 0 to 10, where higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Surgical complications | three months after index surgery
  any complications directly attributable to the surgical intervention
Need for additional treatment | 5 years after index surgery
  rate of patients having to undergo additional surgery / intervention / medication after microvascular decompression
Patient satisfaction | 5yrs after index surgery
  Perceived benefit of surgery as determined by Patient global impression of change (PGIC) scores. The PGIC is a 7-point, patient-reported scale that captures an individual's overall perception of change in their condition. It ranges from "very much improved" to "very much worse," enabling patients to rate whether they feel their health has improved, remained the same, or declined.
Effect of surgical treatment on quality of life | 5 years after index surgery
  Efficacy of microvascular decompression surgery as defined by change of Quality of Life Questionaire as measured by EQ-5D-5L. The EQ-5D-5L is a standardized, patient-reported outcome measure that assesses health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from "no problems" to "extreme problems.

CONTACTS AND LOCATIONS:
Locations (2):
- Dept. of Neurosurgery, RWTH Aachen University Hospital, RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany
- Dept. of Neurosurgery, Cantonal Hospital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided